CLINICAL TRIAL: NCT03717688
Title: The Effects of Neprilysin on Glucagon-like Peptide-1
Acronym: NEP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nicolai Jacob Wewer Albrechtsen (Other)
Responsible Party: Sponsor-Investigator, Nicolai Jacob Wewer Albrechtsen, Junior Consultant, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NEP and GLP-1
Record Dates: First submitted 2018-09-20; First posted 2018-10-24 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Diabetes; Heart Failure
Keywords: GLP-1; Neprilysin; DPP-4
MeSH Terms: conditions — Diabetes Mellitus; Heart Failure | interventions — sacubitril and valsartan sodium hydrate drug combination; Sitagliptin Phosphate; Dipeptidyl-Peptidase IV Inhibitors

STUDY DESIGN:
Intervention Model Description: The participants are on 4 study days with wash out period of minimum 2 weeks randomized to 4 intervention arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo (Placebo Comparator): No treatment. Participants are subjected to a standardized meal
  Interventions: Drug: Placebos
- Entrestro as single dose (Active Comparator): 194 mg sacubitril / 206 mg valstartan (entresto) as one single dose followed by a standardized meal
  Interventions: Drug: Entresto
- Sitagliptin as single dose (Active Comparator): 200mg sitagliptin (100mg the night before and 100mg on the study day) as one single dose followed by a standardized meal
  Interventions: Drug: Sitagliptin 100mg
- Entrestro + sitagliptin as single dose (Active Comparator): 194 mg sacubitril / 206 mg valstartan (entresto) + 200mg sitagliptin (100mg the night before and 100mg on the study day) as one single dose followed by a standardized meal
  Interventions: Drug: Entresto; Drug: Sitagliptin 100mg

INTERVENTIONS:
Drug: Entresto — Single dose administration of Entrestro 194 mg sacubitril / 206 mg valstartan
  Other Names: ARNI; Neprilysin inhibibitor
  Arms: Entrestro + sitagliptin as single dose; Entrestro as single dose
Drug: Sitagliptin 100mg — 2 x 100mg sitagliptin as single dose.
  Other Names: DPP-4 inhibitor
  Arms: Entrestro + sitagliptin as single dose; Sitagliptin as single dose
Drug: Placebos — No treatment
  Other Names: placebo
  Arms: Placebo

SUMMARY:
In the current study we wish to investigate the effects on glucagon-like peptide-1 (GLP-1) of a neprilysin inhibitor

DETAILED DESCRIPTION:
Glucagon-like peptide-1(GLP-1) is secreted during a meal and increases glucose induced insulin secretion. The enzyme dipeptidyl peptidase 4(DPP-4) cleaves intact GLP-1 within minutes and DPP-4 inhibitors are therefore used for treatment of diabetic hyperglycemia. A few animal studies have implicated the enzyme neutral endopeptidase 24.11 (24.11) in the degradation of GLP-1 but if this is the case in humans is unknown. We therefore administered a NEP inhibitor, 194mg sacubitril, a DPP-4 inhibitor (sitagliptin 100mg the night before and 100mg 2 hours before), both, or place, to nine healthy men during a standardized meal and measured plasma concentrations of GLP-1

ELIGIBILITY:
Inclusion Criteria:

* men
* body mass index between 20-25

Exclusion Criteria:

* acute diseases within the two weeks
* chronic diseases
* smoker
* alcoholism, drug addiction or recent weight loss
* blood donation within the last 3 months

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-05-14 (Actual)

PRIMARY OUTCOMES:
GLP-1 | 3 hours after treatment ( during the subsequent standardized meal)
  changes in plasma GLP-1 using immunological methods: intact and total GLP-1

SECONDARY OUTCOMES:
C-peptide | 3 hours after treatment ( during the subsequent standardized meal)
  changes in C-peptide using immunological methods
Glucagon | 3 hours after treatment ( during the subsequent standardized meal)
  Changes in Plasma glucagon concentrations using different analytical methodologies

OTHER OUTCOMES:
Blood glucose | 3 hours after treatment and during the subsequent standardized meal
  changes in blood glucose using immunological methods
GIP | 3 hours after treatment ( during the subsequent standardized meal)
  changes in plasma GIP using immunological methods

CONTACTS AND LOCATIONS:
Locations (1):
- University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
undecided

REFERENCES:
- [Result] Wewer Albrechtsen NJ, Mark PD, Terzic D, Hansen LH, Andersen UO, Hartmann B, Carr RD, Gustafsson F, Deacon CF, Holst JJ, Goetze JP, Plomgaard P. Sacubitril/Valsartan Augments Postprandial Plasma Concentrations of Active GLP-1 When Combined With Sitagliptin in Men. J Clin Endocrinol Metab. 2019 Sep 1;104(9):3868-3876. doi: 10.1210/jc.2019-00515. PMID 31074791
- [Derived] Thonsgaard S, Prickett TCR, Hansen LH, Wewer Albrechtsen NJ, Andersen UO, Terzic D, Plomgaard P, Gustafsson F, Goetze JP, Mark PD. Circulating Concentrations of C-Type Natriuretic Peptides Increase with Sacubitril/Valsartan Treatment in Healthy Young Men. Clin Chem. 2022 May 18;68(5):713-720. doi: 10.1093/clinchem/hvac005. PMID 35175317